CLINICAL TRIAL: NCT03018080
Title: LCI-BRE-H2N-PEPP-001: A Pilot Study of Paclitaxel Plus Pembrolizumab in Patients With Metastatic HER2-Negative Breast Cancer (The PePPy Trial)
Brief Title: Pilot Study of Paclitaxel Plus Pembrolizumab in Metastatic HER2-Negative Breast Cancer
Acronym: PePPy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081370; 00019078 (Other: Advarra IRB); LCI-BRE-H2N-PEPP-001 (Other: Atrium Health)
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Results first posted 2022-10-13 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Breast - Female; Male Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male | interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Phased Pembrolizumab Regimen) (Experimental): Paclitaxel will be given as an IV infusion over 60 minutes, on days 1 and 8 every 21 (+/- 3) days during Cycles 1 and 2. No pembrolizumab will be given during Cycles 1 and 2. Starting with cycle 3 and subsequent cycles, pembrolizumab will be given as an IV infusion over 30 minutes before paclitaxel on day 1 every 21 (+/- 3) days.
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel
- Arm B (Concurrent Pembrolizumab Regimen) (Experimental): Pembrolizumab will be given as an IV infusion on day 1 before paclitaxel every 21 (+/- 3) days. Paclitaxel will be given as an IV infusion over 60 minutes, on days 1 and 8 every 21 (+/- 3) days.
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — IV (in the vein) on day 1 of a 21 day cycle
  Other Names: Keytruda
Drug: Paclitaxel — IV (in the vein) on days 1 and 8 of a 21 day cycle
  Other Names: Taxol

SUMMARY:
The primary objective of this study is to assess the safety and feasibility of the following two regimens: Cohort A) phased regimen of pembrolizumab in which paclitaxel is followed by paclitaxel plus pembrolizumab and Cohort B) concurrent regimen of paclitaxel plus pembrolizumab. The primary safety objective is to evaluate the overall grade 3 or 4 treatment-related adverse event rate for each cohort and compare them to relevant historical controls.

DETAILED DESCRIPTION:
This is an open-label randomized pilot research study to determine if the study drug, pembrolizumab, is safe to use in combination with a chemotherapy drug called paclitaxel. This study will have the following two regimens: Cohort A) phased regimen of pembrolizumab in which paclitaxel is followed by paclitaxel plus pembrolizumab and Cohort B) concurrent regimen of paclitaxel plus pembrolizumab. A total of 40 evaluable subjects will be enrolled over an enrollment period of 18-24 months. The study is planned to enroll approximately 20 evaluable subjects in each treatment cohort.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria:

1. Histologically or cytological confirmed diagnosis of HER2-negative metastatic breast cancer or locally advanced disease not amenable to resection.

   * Available ER and PR status from tumor sample with either hormone receptor positive or negative tumor(s).
   * For subjects with hormone receptor-positive, HER2-negative metastatic breast cancer, they are eligible if they have already received or been intolerant to at least two lines of endocrine therapies (including the adjuvant and/or metastatic setting), or are appropriate candidates for chemotherapy (i.e. large burden of visceral disease).
2. Measurable disease by RECIST 1.1, or evaluable bone disease, i.e., bone lesions that are lytic or mixed (i.e. lytic + sclerotic) in the absence of measurable lesion. Refer to section 11 for the evaluation of measurable disease.
3. Male or female age ≥18 years.
4. ECOG performance status 0, 1 or 2.
5. Must have normal organ and marrow function as defined below:

   * Hematologic - Absolute neutrophil count ≥1,500/mcL

     - Platelets ≥75,000/mcL

     - Hemoglobin ≥ 9 g/dL
   * Renal

     * Creatinine ≤ 1.5X ULN or
     * Measured or calculated creatinine clearance (CrCl) ≥ 30 mL/min for subject with creatinine levels > 1.5X ULN [CrCl should be calculated per institutional standard; GFR can also be used in place of creatinine or CrCl]
   * Hepatic

     * Total bilirubin ≤1.5X ULN or for subjects with total bilirubin levels >1.5X ULN, direct bilirubin ≤ULN
     * AST(SGOT)/ALT(SGPT) ≤2.5X ULN
   * Coagulation

     * PT and PTT ≤ 1.5X ULN; subjects receiving anticoagulant therapy are eligible if PT or PTT is within therapeutic range of intended use of anticoagulants per investigator discretion.
     * INR ≤ 1.5; Patients receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation per investigator discretion.
6. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to receiving C1D1.
7. Female subjects of childbearing potential must be willing to use an adequate method of birth control as outlined in Section 8.1.10, be surgically sterile, or abstain from heterosexual activity for the course of the study and 120 days after the last dose of study therapy. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Male subjects of reproductive potential should agree to use an adequate method of contraception starting with the first dose of study therapy and 120 days after the last dose of study therapy. Abstinence is acceptable if this is the established and preferred contraception for the subject.
8. Has completed the screening requirement of a core or punch biopsy of a tumor lesion per Section 5 (bone tissue not acceptable). Biopsy of the breast tumor or other regional areas is acceptable (i.e. lymph nodes, skin lesions).

   * Subjects who are unable to meet the screening requirement of a tumor biopsy due to inaccessible tumor, subject safety concern, or bone-only disease may submit an archived tumor specimen from primary tumor or metastatic biopsy collected within 12 months from consent.
   * Subjects who decline tumor biopsy may submit archived tumor specimen as specified above (within 12 months from consent) only after Sponsor-Investigator approval.
9. Ability to understand and the willingness to sign the written informed consent document.

Exclusion Criteria

Subjects must not meet any of the following criteria:

1. Prior chemotherapy within 3 weeks, prior targeted small molecule therapy or radiation therapy within 2 weeks, or prior anti-cancer monoclonal antibody (mAb) for direct anti-neoplastic treatment within 4 weeks prior to Cycle 1 Day 1.
2. Not recovered (i.e., ≤ Grade 1) from adverse events due to agents previously administered.

   o Note: Subjects with ≤ Grade 2 neuropathy or alopecia of any grade are an exception and may qualify for the study.
3. More than three prior lines of chemotherapy for HER2-negative metastatic disease or for locally advanced disease that is not amenable to resection.

   o Note: Non-Chemotherapy regimens do not count as prior lines (ex: hormonals, biologics)
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137) or has participated in Merck MK-3475 trial(s) and received MK-3475 as part of protocol therapy.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Cycle 1 Day 1
6. Has had major surgery within 3 weeks prior to Cycle 1 Day 1.
7. Has received any other investigational agents within 4 weeks of Cycle 1 Day 1 of study therapy.
8. Known active uncontrolled or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis as indicated by clinical symptoms, cerebral edema, and/or progressive growth.

   o Note: Subjects with treated CNS metastases are eligible if they are asymptomatic, have no requirement for steroids, no requirement for anticonvulsants, and stable CNS radiographic study showing no significant vasogenic edema ≥ 4 weeks since completion of radiation and ≥ 2 weeks since discontinuation of steroids.
9. History of known allergic reaction to paclitaxel
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment. Pregnant women are excluded from this study because paclitaxel is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with paclitaxel, breastfeeding should be discontinued if the mother is treated with paclitaxel. These potential risks also apply to pembrolizumab being used in this study.
12. Has a known history of Human Immunodeficiency Virus (HIV) or known acquired immunodeficiency disorder (AIDS). HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with paclitaxel and pembrolizumab. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
13. Has known active infection with hepatitis B or hepatitis C.
14. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

    o Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has a known additional malignancy that progressed or required active treatment within the last 5 years.

    o Note: Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
16. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
17. Has an active infection requiring systemic therapy.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Has received a live vaccine within 30 days of Cycle 1 Day 1 of study therapy. o Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Tan, MD, Principal Investigator — Atrium Health (formerly Carolinas HealthCare System)
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nanda R, Chow LQ, Dees EC, Berger R, Gupta S, Geva R, Pusztai L, Pathiraja K, Aktan G, Cheng JD, Karantza V, Buisseret L. Pembrolizumab in Patients With Advanced Triple-Negative Breast Cancer: Phase Ib KEYNOTE-012 Study. J Clin Oncol. 2016 Jul 20;34(21):2460-7. doi: 10.1200/JCO.2015.64.8931. Epub 2016 May 2. PMID 27138582
- [Result] Tan AR, Chai SJ, Robinson MM, Hellner LB, Gavini N, Sulai N, Turner JD, Atlas J, Graham DL, Induru RR, Kadakia KC, Vallabhanei GD, Heeke AL, Foureau DM, Fisher JG. A pilot study of paclitaxel plus pembrolizumab in patients with metastatic HER2-negative breast cancer (PePPy). Cancer Research. 2022; 82(4_Supplement): P2-14-03

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen)
Started | 21 | 19
Completed | 9 | 0
Not Completed | 12 | 19
Not completed — Death | 12 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen) | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 6 | 7 | 13
Age, Continuous [Median (Full Range); unit: years] | 54 [28 to 73] | 57 [40 to 76] | 56.5 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40
ECOG at Baseline [Count of Participants; unit: Participants] — Measure Description: ECOG Scale of Performance Status, developed by the Eastern Cooperative Oncology Group.
  (0) subject is fully active, able to carry on all predisease performance without restriction; (1) subject is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light house work, office work); (2) subject is ambulatory and capable of all self-care but unable to carry out any work activities (up and about more than 50% of waking hours)
  Participants
    0 | 12 | 5 | 17
    1 | 8 | 13 | 21
    2 | 1 | 1 | 2
Hormone Receptor Status [Count of Participants; unit: Participants] — Hormone receptor (HR) status was determined based on tumor samples. Subject was HR positive if ER% or PR% were >=10%. If ER% and PR% were <10%, then subject was considered HR negative.
  Participants
    HR Positive | 10 | 10 | 20
    HR Negative | 11 | 9 | 20
Prior Paclitaxel Exposure [Count of Participants; unit: Participants] — Indicates whether or not the subject had previously received paclitaxel in any setting.
  Participants
    Prior Paclitaxel | 9 | 5 | 14
    No Prior Paclitaxel | 11 | 12 | 23
    Unknown | 1 | 2 | 3
Prior Docetaxel Exposure [Count of Participants; unit: Participants] — Indicates whether or not the subject had previously received docetaxel in any setting
  Participants
    Prior Docetaxel | 6 | 12 | 18
    No Prior Docetaxel | 14 | 6 | 20
    Unknown | 1 | 1 | 2
Number of Prior Metastatic Chemotherapy Lines [Count of Participants; unit: Participants] — Indicates the number of prior lines of chemotherapy that the subject received in the metastatic setting
  Participants
    0 | 12 | 6 | 18
    1 | 7 | 6 | 13
    2 | 2 | 6 | 8
    3 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Grade 3 or 4 Treatment-related Adverse Event
Description: Grade 3 or 4 study treatment-related adverse events will be determined for each subject as a binary variable indicating whether or not the subject experienced at least one grade 3 or 4 study treatment-related adverse events according to the NCI Common Terminology for Adverse Events, version 4.0. An adverse event will be considered study treatment related if it is determined that the event is at least possibly related to either paclitaxel, pembrolizumab, or both.
Time Frame: From enrollment to at least 30 days following cessation of study treatment. The median time on treatment was 5.5 months.
Population: The evaluable population will consist of all randomized subjects who begin study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen)
Number analyzed (Participants) | 21 | 19
Participants | 5 | 6
Statistical Analysis 1: Comparison: Arm A (Phased Pembrolizumab Regimen); The reported grade 3/4 toxicity rate with weekly paclitaxel was 0.35. If it became evident that the grade 3/4 treatment-related toxicity rate on either arm convincingly exceeded 0.35, the study arm would have been halted. Convincing evidence of exceeding 0.35 was based on Bayesian methods and continuous monitoring, where the stopping rule would have held enrollment if the posterior probability at any point exceeded 0.50 or higher; Test type: Other — Estimation only; Rate = 0.238, 95% CI 2-sided [0.082 to 0.472] — Confidence interval estimated using the Clopper Pearson method
Statistical Analysis 2: Comparison: Arm B (Concurrent Pembrolizumab Regimen); [analysis description as in outcome 1, analysis 1]; Test type: Other — Estimation only; Rate = 0.316, 95% CI 2-sided [0.126 to 0.566] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Number of Subjects With an Objective Response (Per RECIST V1.1)
Description: Objective response was determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of complete response (CR) or partial response (PR) as determined by RECIST 1.1 response criteria. A CR is indicated by disappearance of all target and non target lesions. A PR is indicated by >=30% decrease in sum of longest diameter of target lesions with baseline as reference.
Time Frame: From enrollment to best response while on study treatment; subjects remained on treatment until disease progression or death or unacceptable toxicity (subjects were on treatment for a median of 5.5 months)
Population: The evaluable population will consist of all randomized subjects who begin study therapy and have measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen)
Number analyzed (Participants) | 21 | 19
Participants | 4 | 8
Statistical Analysis 1: Comparison: Arm A (Phased Pembrolizumab Regimen); Test type: Other — Estimation only; Rate = 0.191, 95% CI 2-sided [0.055 to 0.419] — Confidence interval estimated using the Clopper Pearson method
Statistical Analysis 2: Comparison: Arm B (Concurrent Pembrolizumab Regimen); Test type: Other — Estimation only; Rate = 0.421, 95% CI 2-sided [0.203 to 0.665] — Confidence interval estimated using the Clopper Pearson method

3. Secondary Outcome: Progression-free Survival (PFS) Per RECIST 1.1
Description: PFS is defined as the duration of time from treatment start date to first occurrence of either progressive disease (PD) or death. PD must be objectively determined per RECIST 1.1 criteria, where progression date is date of last assessment that identified PD. If subject died without documented PD, progression date will be death date. For surviving subjects who do not have PD, PFS will be censored at the date of last disease assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, PFS will be censored at the date of last disease assessment prior to commencement of subsequent therapy. Subjects who have an initial PFS event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Time Frame: From treatment start date to date of progression/death, or censored as described; assessed for approximately 2 years.
Population: The evaluable population for PFS consisted of all randomized subjects who begin study therapy
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen)
Number analyzed (Participants) | 21 | 19
Months | 4.1 [1.4 to 6.9] | 3.9 [1.4 to 6.8]
Statistical Analysis 1: Comparison: Arm A (Phased Pembrolizumab Regimen); Test type: Other — Estimation only; Median = 4.1, 95% CI 2-sided [1.4 to 6.9] — The Kaplan Meier method was used to estimate the median PFS(in months) for the population. The Greenwood method was used to estimate the confidence limits of the median progression free survival
Statistical Analysis 2: Comparison: Arm B (Concurrent Pembrolizumab Regimen); Test type: Other — Estimation only; Median = 3.9, 95% CI 2-sided [1.4 to 6.8] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration from treatment start date to the date of death from any cause. Subjects who are alive or lost to follow up at the time of the analysis will be censored at the last known date they were alive.
Time Frame: From date of treatment start to date of death, or censored as described; assessed for approximately 5 years.
Population: The evaluable population consisted of all randomized subjects who begin study therapy.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen)
Number analyzed (Participants) | 21 | 19
Months | 27.6 [9.7 to NA] — Upper limit of the confidence interval is not reached due to censoring rate | 9.0 [6.8 to 14.0]
Statistical Analysis 1: Comparison: Arm A (Phased Pembrolizumab Regimen); Test type: Other — Estimation only; Median = 27.6, 95% CI 2-sided [lower limit 9.7] (Upper limit of the confidence interval is not reached due to censoring rate) — The Kaplan Meier method was used to estimate median OS (in months). The Greenwood method was used to estimate confidence limits of median overall survival
Statistical Analysis 2: Comparison: Arm B (Concurrent Pembrolizumab Regimen); Test type: Other — Estimation only; Median = 9.0, 95% CI 2-sided [6.8 to 14.0] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Number of Subjects With Disease Control (Per RECIST V1.1)
Description: Disease control was determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of complete response (CR), partial response (PR), or stable disease (SD) as determined by RECIST 1.1 response criteria. A CR is indicated by disappearance of all target and non target lesions. A PR is indicated by >=30% decrease in sum of longest diameter of target lesions with baseline as reference. SD is indicated by neither sufficient shrinkage to qualify for PR nor sufficient growth from nadir (>=20%) to indicate progression.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen)
Number analyzed (Participants) | 21 | 19
Participants | 14 | 12
Statistical Analysis 1: Comparison: Arm A (Phased Pembrolizumab Regimen); Test type: Other — Estimation only; Rate = 0.667, 95% CI 2-sided [0.430 to 0.854] — Confidence interval estimated using the Clopper Pearson method
Statistical Analysis 2: Comparison: Arm B (Concurrent Pembrolizumab Regimen); Test type: Other — Estimation only; Rate = 0.632, 95% CI 2-sided [0.384 to 0.837] — Confidence interval estimated using the Clopper Pearson method

6. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) is defined as the duration of time from the first assessment that determined a CR or PR to the date of the first occurrence of progressive disease or death. Progression events and the censoring mechanism for DoR will be the same as described for PFS. DoR will be determined for each subject using the RECIST 1.1 criteria.
Time Frame: From date of response to date of progression/death, or censored as described above; assessed for approximately 2 years.
Population: The evaluable population consisted of all randomized subjects who begin study therapy and achieve objective response (CR or PR) on study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen)
Number analyzed (Participants) | 4 | 8
Months | 7.3 [5.6 to 8.3] | 4.0 [2.6 to 8.3]
Statistical Analysis 1: Comparison: Arm A (Phased Pembrolizumab Regimen); Test type: Other — Estimation only; Median = 7.3, 95% CI 2-sided [5.6 to 8.3] — The Kaplan Meier method was used to estimate median duration of response (in months). The Greenwood method was used to estimate confidence limits of median duration of response
Statistical Analysis 2: Comparison: Arm B (Concurrent Pembrolizumab Regimen); Test type: Other — Estimation only; Median = 4.0, 95% CI 2-sided [2.6 to 8.3] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline, during treatment, and through 30 days after study treatment is discontinued, an average of 14 months.
Arm/Group | Arm A (Phased Pembrolizumab Regimen) | Arm B (Concurrent Pembrolizumab Regimen)
All-Cause Mortality (participants affected / at risk) | 12/21 | 19/19
Serious Adverse Events (participants affected / at risk) | 4/21 | 7/19
Other Adverse Events (participants affected / at risk) | 21/21 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Phased Pembrolizumab Regimen) (N=21) | Arm B (Concurrent Pembrolizumab Regimen) (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 — Gastroenteritis
Death NOS (General disorders) | 0 | 2
Fever (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Skin infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Phased Pembrolizumab Regimen) (N=21) | Arm B (Concurrent Pembrolizumab Regimen) (N=19)
Anemia (Blood and lymphatic system disorders) | 3 | 5
Atrial flutter (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 6 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 1 | 0 — intermittent R eye sty
Flashing lights (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Bloating (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 5 | 5
Diarrhea (Gastrointestinal disorders) | 4 | 7
Dry mouth (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1 — Diverticulitis
Mucositis oral (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 7 | 8
Vomiting (Gastrointestinal disorders) | 2 | 6
Chills (General disorders) | 2 | 1
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 3 | 3
Fatigue (General disorders) | 15 | 11
Fever (General disorders) | 1 | 2
Gait disturbance (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 4 | 2
Localized edema (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 6 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 0 — cholangitis
Allergic reaction (Immune system disorders) | 1 | 0
Breast infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 0 — SHINGLES
Laryngitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Lymph gland infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 1
Nail infection (Infections and infestations) | 1 | 0
Papulopustular rash (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 3 | 0
Skin infection (Infections and infestations) | 2 | 1
Upper respiratory infection (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 1 | 2
Vaginal infection (Infections and infestations) | 0 | 1
Vulval infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Alkaline phosphatase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 1 | 0
Serum amylase increased (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 | 0 — Vit B12 deficiency
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 1 — L jaw
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 1 — restless leg
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Dizziness (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 8 | 4
Paresthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 13
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 2 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Chest congestion
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 2
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0 — dermatitis
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 — foreign body reaction
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 — ingrown toenail
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1 — acne
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1 — generalized rash
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 1
Hot flashes (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Lymphedema (Vascular disorders) | 2 | 0
Thromboembolic event (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT03018080/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT03018080/ICF_001.pdf